CLINICAL TRIAL: NCT00578734
Title: A Multicenter, Randomized, Masked, Placebo-Controlled Trial to Assess the Safety and Efficacy of Lucinactant in Acute Hypoxemic Respiratory Failure in Children Up to Two Years of Age
Brief Title: Lucinactant for Treatment of Acute Hypoxemic Respiratory Failure in Children up to Two Years Old
Acronym: KL4-AHRF-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Windtree Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KL4-AHRF-01
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Results first posted 2012-04-27 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Acute Hypoxemic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — lucinactant; Surface-Active Agents

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lucinactant (Experimental): SURFAXIN® (lucinactant) for intratracheal instillation
  Interventions: Drug: Lucinactant
- Sham Air (Sham Comparator): Sham air (placebo) instillation
  Interventions: Other: Sham Comparator

INTERVENTIONS:
Drug: Lucinactant — Slow intra-tracheal instillation
  Other Names: SURFAXIN®; Surfactant
  Arms: Lucinactant
Other: Sham Comparator — Slow intra-tracheal instillation
  Other Names: Placebo
  Arms: Sham Air

SUMMARY:
Treatment with lucinactant, a peptide-containing synthetic lung surfactant, will be evaluated in young children with acute respiratory failure who require mechanical ventilation (life support), to determine if it is safe and if treatment with lucinactant will reduce the number of days a child needs mechanical ventilation (life support).

DETAILED DESCRIPTION:
Determine the safety and tolerability of administration of a peptide-containing synthetic lung surfactant, lucinactant, in children up to two years of age and assess whether treatment with lucinactant can decrease the duration of mechanical ventilation in young children.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 38 weeks (corrected age) to 2 years (24 months)
* Intubated and mechanically ventilated (MV) for ≥ 6 hours and anticipated need for MV for ≥ 24 hours
* Persistent hypoxia
* Written informed consent

Exclusion Criteria:

* Mechanical Ventilation for > 48 hours
* Oxygenation index ≥ 25, if arterial line was avialable
* Pre-existing clinically significant or palliated/uncorrected cardiac disease adversely affecting cardiopulmonary function and gas exchange
* Neuromuscular disease or hypotonia
* Upper airway disease
* Baseline requirment for supplemental oxygen
* Untreated pneumothorax
* Off-label use of commercially available surfactant outside neonatal period
* History of prematurity and passive immunoprophylaxis with humanized monoclonal antibody
* Head injury with Glasgow Coma Scale < 8
* Brain death or impending brain death
* Do not resuscitate orders
* Cardiopulmonary resuscitation within 6 hours of meeting entry criteria
* Experimental therapy in which the intervention potentially affects respiratory outcomes
* Any transplant recipient
* Meconium aspiration syndrome
* Bordetella pertussis infection confirmed via laboratory tests and/or highly suspected pertussis infection

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 165 (Actual)
Dates: Start 2007-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Thomas, MD, Principal Investigator — Milton S. Hershey Medical Center; Adrienne Randolph, MD, Principal Investigator — Boston Children's Hospital
Locations (3):
- Call for information, Warrington, Pennsylvania, United States
- Chile (2):
  - Call for Information, Concepción
  - Call For Information, Santiago

REFERENCES:
- [Derived] Thomas NJ, Guardia CG, Moya FR, Cheifetz IM, Markovitz B, Cruces P, Barton P, Segal R, Simmons P, Randolph AG; PALISI Network. A pilot, randomized, controlled clinical trial of lucinactant, a peptide-containing synthetic surfactant, in infants with acute hypoxemic respiratory failure. Pediatr Crit Care Med. 2012 Nov;13(6):646-53. doi: 10.1097/PCC.0b013e3182517bec. PMID 22791092

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 24 hospitals in the United States and Chile from 04 June, 2007 to 23 March, 2010. Last subject's last visit occurred on 05 April, 2010.
Groups:
- Lucinactant: KL₄Surfactant (lucinactant) endotracheal instillation
Period: Overall Study
Arm/Group | Lucinactant | Sham Air
Started | 84 | 81
Completed | 84 | 81
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lucinactant | Sham Air | Total
Number analyzed (Participants) | 84 | 81 | 165
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 84 | 81 | 165
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 0.44 (0.43) | 0.45 (0.43) | 0.45 (0.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 27 | 56
  Male | 55 | 54 | 109
Region of Enrollment [Number; unit: participants]
  United States | 28 | 27 | 55
  Chile | 56 | 54 | 110

OUTCOME MEASURES:

1. Primary Outcome: Duration of Mechanical Ventilation Through 14 Days
Description: Duration of mechanical ventilation (MV) from baseline to successful extubation (not receiving MV for at least 24 hours) through a maximum of 14 days.
Time Frame: Up to 14 Days
Population: The sample size calculation was based on historical data and expected treatment effect. The primary efficacy analysis was for the intent-to-treat population, defined as all randomized subjects (N=165). A supportive population (N=134) of subjects without a major protocol violation that could impact efficacy was also used for efficacy analyses.
Measure: Least Squares Mean (95% Confidence Interval); unit: days
Arm/Group | Lucinactant | Sham Air
Number analyzed (Participants) | 84 | 81
days | 4.0 [3.5 to 4.6] | 4.5 [3.9 to 5.2]

2. Secondary Outcome: Ventilator-free Days; Duration of Days on Oxygen, Intensive Care Unit (ICU) Stay, and Hospitalization Through 14 Days
Time Frame: Up to 14 days
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: days
Arm/Group | Lucinactant | Sham Air
Number analyzed (Participants) | 84 | 81
days
  Ventilator-free days | 5.2 [4.6 to 5.9] | 4.6 [4.1 to 5.3]
  Duration in Pediatric Intensive Care Unit (PICU) | 6.2 [5.4 to 7.0] | 6.7 [5.9 to 7.6]
  Duration of Supplemental Oxygen | 7.7 [6.8 to 8.7] | 7.9 [7.0 to 9.0]
  Duration of Hospitalization | 10.0 [9.1 to 11.1] | 9.7 [8.8 to 10.7]

ADVERSE EVENTS:
Time Frame: 14 days from randomization or until resolution of adverse events.
Arm/Group | Lucinactant | Sham Air
Serious Adverse Events (participants affected / at risk) | 20/84 | 14/81
Other Adverse Events (participants affected / at risk) | 65/84 | 62/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lucinactant (N=84) | Sham Air (N=81)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (2)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Coarctation of the aorta (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Oxygen saturation decreased (Investigations) | 2 (2) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Neurological symptom (Nervous system disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pertussis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lucinactant (N=84) | Sham Air (N=81)
Anaemia (Blood and lymphatic system disorders) | 11 (13) | 19 (21)
Bradycardia (Cardiac disorders) | 4 (4) | 9 (10)
Abdominal distension (Gastrointestinal disorders) | 5 (5) | 3 (3)
Drug withdrawal syndrome (General disorders) | 4 (4) | 4 (4)
Oedema (General disorders) | 2 (2) | 5 (6)
Pyrexia (General disorders) | 2 (2) | 4 (4)
Pneumonia (Infections and infestations) | 7 (7) | 2 (2)
Oxygen saturation decreased (Investigations) | 9 (10) | 6 (10)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 12 (12) | 6 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 6 (6) | 6 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 23 (23) | 17 (18)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 4 (5)
Metabolic alkalosis (Metabolism and nutrition disorders) | 5 (5) | 9 (9)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 13 (13)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 5 (5)
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (5)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (7)
Stridor (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (10)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Capillary leak syndrome (Vascular disorders) | 4 (4) | 3 (3)
Hypertension (Vascular disorders) | 5 (5) | 3 (3)
Hypotension (Vascular disorders) | 8 (8) | 12 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
First publication must be joint, multicenter publication in conjunction with a presentation. Following multicenter publication, proposed publications or presentations must be submitted to sponsor 30 days in advance. In the event of an objection by sponsor, PI agrees to delay the publication or presentation until modifications or revisions have been made to protect Sponsor's patent rights, copyrights, or proprietary rights.